CLINICAL TRIAL: NCT05789602
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BPI-460372 in Advanced Solid Tumor Patients
Brief Title: A Study of BPI-460372 in Advanced Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661911
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Oral tablets taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with BPI-460372 administered, once daily (QD).
  Interventions: Drug: BPI-460372
- Dose Expansion (Experimental): Oral tablets administered at MTD/RP2D defined dose. Each treatment cycle will be 21 days in duration with BPI-460372 administered, once daily (QD)
  Interventions: Drug: BPI-460372

INTERVENTIONS:
Drug: BPI-460372 — Subjects will receive BPI-460372 until disease progression

SUMMARY:
This study is an open-label, single arm, dose escalation and dose expansion phase 1 study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of BPI-460372 in solid tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18, male and female patients；
* Expected survival ≥ 3 months；
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Dose escalation phase: histologically or cytologically confirmed locally advanced or metastatic solid tumor patients, who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Dose expansion phase: histologically or cytologically confirmed locally advanced Malignant mesothelioma, Epithelioid hemangioendothelioma or other diagnosed solid tumor patients with NF2 defects, YAP/TAZ fusion, LATS1/2 mutations, and other Hippo signaling pathway abnormalities , who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Evaluable lesion required for dose escalation phase and at least 1 measurable lesion as per RECIST v1.1 or mRECIST v1.1 required for dose expansion phase;

Exclusion Criteria:

* Patients who have previously received a TEAD inhibitor;
* Inadequate wash-out of prior therapies described per protocol, which may include anti-tumor therapies, tumor adjuvant drugs, organ or stem cell transplantation，etc；
* Patients with severe or unstable systemic disease, unstable/symptomatic CNS metastasis, meningeal metastasis and spinal cord compression，malignant tumors, cardiac disease, bleeding or embolic disease, infectious disease, conditions affecting drug swallow and absorption, medical history leading to chronic diarrhea, etc;
* Pregnancy or lactation;
* Other conditions considered not appropriate to participate in this trial by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
The adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
The dose-limiting toxicity（DLT） | Through the Phase I, approximately 24 months
  The dose-limiting toxicity
Determine the Maximum Tolerated Dose (MTD) | Through the Phase I, approximately 24 months
  The MTD will be based on DLT.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of BPI-460372 | Time Frame: Through the Phase I, approximately 24 months
  Based on blood plasma concentration
Evaluate the effectiveness of BPI-460372 | Time Frame: Through the Phase I, approximately 24 months
  Efficacy assessments (tumor evaluation) will be performed per RECIST1.1 or mRECIST1.1

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Zhengzhou

IPD SHARING:
Plan to Share IPD: No